CLINICAL TRIAL: NCT01032278
Title: A Multicenter Study in Patients Undergoing AnthRacycline-Based Chemotherapy to Assess the Effectiveness of Using Biomarkers to Detect and Identify Cardiotoxicity and Describe Treatment (PREDICT)
Brief Title: Effectiveness of Using Biomarkers to Detect and Identify Cardiotoxicity and Describe Treatment (PREDICT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Alere San Diego (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000660615; MDA-2007-0914A; CDR0000660615 (Other: NCI Clinical Trials); NCI-2011-01466 (Registry Identifier: NCI CTRP); NCT01311843 (obsolete NCT alias)
Record Dates: First submitted 2009-12-13; First posted 2009-12-15 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Toxicity; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: cardiac toxicity; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Cardiotoxicity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Biomarker Testing (Experimental): Biomarker testing for cardiac biomarkers, B-type natriuretic peptide (BNP) and Troponin I (TnI), and symptom questionnaires of participants undergoing anthracycline-based chemotherapy.
  Interventions: Other: Laboratory Biomarker Analysis; Behavioral: Questionnaires

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Blood drawn for biomarker analysis at baseline, before each chemotherapy visit, 6 months after starting chemotherapy, and 12 months after completion of chemotherapy.
  Other Names: Biomarker Testing
Behavioral: Questionnaires — Symptom questionnaire completion at baseline, beginning of every third cycle of chemotherapy, 6 months after starting chemotherapy, and 12 months after completion of chemotherapy.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to learn if certain biomarker testing on blood samples can help to detect heart damage that may occur during chemotherapy. Biomarkers are chemical "markers" found in the blood that may be related to heart function. High levels of these markers may be linked with heart problems such as heart damage.

DETAILED DESCRIPTION:
Study Visits:

If you are found to be eligible to take part in this study, you will have study tests and procedures performed on the same days as your visits for chemotherapy treatment. These study visits will occur about every 3-4 weeks apart. The exact number and timing of the visits will depend on when your scheduled chemotherapy visits occur. You and your doctor will discuss the best chemotherapy treatment and schedule for you.

At each chemotherapy visit, before you receive your chemotherapy the following tests and procedures will be performed:

* You will have a physical exam, including measurement of vital signs.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* Additional blood (about 1 teaspoon) will be drawn for biomarker testing.

At the beginning of every third cycle of chemotherapy you will be asked to complete a questionnaire about any symptoms you may be experiencing.

Follow-Up Visit:

At about 6 months after starting your chemotherapy the following tests and procedures will be performed:

* You will complete the symptom questionnaire.
* You will have a physical exam, including measurement of vital signs.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* Additional blood (about 1 teaspoon) will be drawn for biomarker testing.
* You will have an ECG.
* You will have an ECHO or MUGA scan.

End-of-Study Visit:

At about 12 months after starting your chemotherapy you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will complete the symptom questionnaire.
* You will have a physical exam, including measurement of vital signs.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* Additional blood (about 1 teaspoon) will be drawn for biomarker testing.
* You will have an ECG.
* You will have an ECHO or MUGA scan.

At any time during the study, if your doctor thinks it is necessary, you will have an ECG and/or ECHO or MUGA scan.

If you stop receiving chemotherapy during your participation in this study, you will still be asked to complete the above tests and procedures listed at the 12-month (end-of-study visit) visit. Other tests and procedures scheduled during the study may not be performed because you are no longer receiving chemotherapy treatment. Your study doctor and the research staff will go over this information with you if this happens.

Research Test Results:

The primary biomarkers being tested in this study are the BNP and TnI. Both the BNP and TnI look at the function of your heart. The BNP and TnI will both be tested at MD Anderson.

The results of the biomarker tests will be kept separately from your other tests results, and will not affect your treatment in any way. The only reason your biomarker test results would be shared with your cancer doctor would be if the study doctor thinks the results show a heart problem. In that case, the study doctor will contact you right away to advise you about what to do next (for example, coming in to the clinic). You will be referred to a cardiologist (heart doctor) if the study doctor decides it is necessary.

In addition to the biomarkers being tested in this study, if you had ECHOs during the study, the images of the ECHOs may be copied to a DVD and sent to the University of Pennsylvania for review related to research on heart damage caused by anthracycline-based chemotherapy. Before sending your ECHOs to the University of Pennsylvania MD Anderson will remove all of your personal identifiers (name, date of birth, age, and medical record number) included on the ECHO imaging DVD.

Length of Study Participation:

Your study participation will last about 12 months from date of your first chemotherapy treatment. You will have a follow up visit at about 6 months from the date of your first chemotherapy and an end of study visit at about 12 months from the date of your first chemotherapy treatment. This will end your participation in the study.

This is an investigational study. At this time, the biomarker testing in this study is only being used in research. Its use in detecting heart damage is considered investigational.

Up to 830 patients will take part in this multicenter study. Up to 200 will be enrolled at the Harris Health System and MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 18 years or older
2. Starting a new course of chemotherapy that includes an anthracycline (does not have to be first-line therapy and previous anthracycline use is allowed)
3. Has a life expectancy greater than 12 months

Exclusion Criteria:

1. Unstable angina within the last 3 months of registration
2. Myocardial infarction within the last 3 months of registration
3. LVEF less than 50%
4. Patients receiving concurrent dexrazoxane
5. Decompensated Heart Failure in the last 3 months prior to registration
6. Prior symptomatic arrhythmia (within 3 months of study registration)
7. Severe pulmonary disease (FEV </= 1.0 liters), and/or pulmonary hypertension (mean pulmonary artery pressure >/=60mm Hg), and/or dependent use of oxygen
8. BNP >/= 200 pg/ml or BNP >/= 200 pg/ml and troponin I >/= 0.4 ng/ml via use of the Biosite Triage Profiler Note: BNP or BNP and TnI resulted in a local lab within 30 days of starting anthracycline based chemotherapy may be used in determining eligibility. Results, either by the Biosite Triage Profiler or the local lab, > /= the parameters described in exclusion 3.2.8 deem the patient ineligible for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2011-01-25 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Use of Cardiac Biomarkers, B-type Natriuretic Peptide (BNP) and Troponin I (TnI), for Detecting Cardiotoxicity in Patients Undergoing Anthracycline-based Chemotherapy | 12 months
  Cardiotoxicity defined as presentation of one or more cardiac events within 12 months of initiation of chemotherapy. Cardiac event defined as any new symptomatic cardiac arrhythmia, acute coronary syndrome, symptomatic HF, development of asymptomatic left ventricular dysfunction (defined as left ventricular ejection fraction (LVEF) reduction of 10% to less than 50% or a decrease of greater than 15% from baseline), or sudden cardiac death (defined as rapid and unexpected death from cardiac causes with or without known underlying heart disease). BNP greater than 200 pg/ml is considered abnormal. Troponin I greater than 0.4 ng/ml is also considered abnormal. Patients having at least one abnormal evaluation preceding cardiotoxicity for either biomarker (i.e., one abnormal troponin or one abnormal BNP assessments) classified as having an abnormal test.
  Primary analysis performed using data from all subjects with at least one post baseline biomarker measure for BNP and/or troponin I.

SECONDARY OUTCOMES:
Sensitivity and specificity of serial LVEF measurements in detecting cardiotoxicity | 12 months
Clinical management and outcomes of patients with abnormal cardiac biomarkers or clinically defined cardiotoxicity during chemotherapy | 12 months
Supportive utility of patient-reported symptoms for the development of cardiac-related toxicity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Wolff, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon B. Johnson General Hospital (LBJ), Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Narayan HK, Wei W, Feng Z, Lenihan D, Plappert T, Englefield V, Fisch M, Ky B. Cardiac mechanics and dysfunction with anthracyclines in the community: results from the PREDICT study. Open Heart. 2017 Jan 16;4(1):e000524. doi: 10.1136/openhrt-2016-000524. eCollection 2017. PMID 28123764
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org